CLINICAL TRIAL: NCT03754595
Title: Application of 2D and 3D Laparoscopy in Laparoscopic Pancreaticoduodenectomy: a Prospective Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DaiMH
Record Dates: First submitted 2018-11-25; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Pancreatoduodenectomy
Keywords: 2D and 3D Laparoscopic pancreatoduodenectomy

STUDY DESIGN:
Intervention Model Description: Two parallel groups: 2DLaparoscopic pancreatoduodenectomy and 3DLaparoscopic pancreatoduodenectomy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2D Laparoscopic pancreatoduodenectomy (Active Comparator): Patients with pancreatic cancer treated by 2D Laparoscopic pancreatoduodenectomy
  Interventions: Procedure: 2D Laparoscopic pancreatoduodenectomy
- 3D Laparoscopic pancreatoduodenectomy (Experimental): Patients with pancreatic cancer treated by 3D Laparoscopic pancreatoduodenectomy
  Interventions: Procedure: 3D Laparoscopic pancreatoduodenectomy

INTERVENTIONS:
Procedure: 3D Laparoscopic pancreatoduodenectomy — Patients with pancreatic cancer treated by 3D Laparoscopic pancreatoduodenectomy
  Arms: 3D Laparoscopic pancreatoduodenectomy
Procedure: 2D Laparoscopic pancreatoduodenectomy — 2D Laparoscopic pancreatoduodenectomy
  Arms: 2D Laparoscopic pancreatoduodenectomy

SUMMARY:
Pancreatic cancer is extremely malignant, with a low sensibility to chemotherapy and radiotherapy, and a poor prognosis. Surgical treatment is very important for pancreatic cancer. Laparoscopic pancreatoduodenectomy is a standard radical procedure we are going to compare and discuss the advantages of 2D and 3D Laparoscopic pancreatoduodenectomy in our RCT study.

DETAILED DESCRIPTION:
This study is to compare the efficiency and safety between 2D laparoscopic pancreatoduodenectomy and 2D laparoscopic pancreaticoduodenectomy for pancreatic cancer. We design a prospective randomized study. Patients with malignant pancreatic tumor who underwent pancreatoduodenectomy are recruited to the study. After obtaining informed consent, eligible patients are randomly allocated to 2D laparoscopic or 3D laparoscopic group before the operation day . The outcomes evaluated were hospital stay, and blood loss, radicality of surgery, duration of operation and complication rate.

ELIGIBILITY:
Inclusion Criteria:

Age: >18yr, <75yr Patients with pancreatic cancer or non-pancreatic cancers (biliary duct cancer or ampullary cancer) who underwent pancreatoduodenectomy Preoperative imaging assessment is resectable or borderline resectable -

Exclusion Criteria:

- Benign tumors of the head of pancreas Enhanced CT diagnosis revealed that the excess of SMV was more than 180 degrees, or distant metastasis.

conversion to laparotomy because of intraoperative difficulty

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 60 month
  overall survival duration after surgical treatment

SECONDARY OUTCOMES:
Overall complications | Up to postoperative 30 days
  The proportion of all complications after operation accounted for the total number of patients

OTHER OUTCOMES:
Operative time | 12 hours
  Durtion of operation
Pancreatic fistula | Up to postoperative 30 days
  The international study group (ISGPF) definition: A drain output of any measurable volume of fluid on or after postoperative day 3 with an amylase content greater than 3 times the serum amylase activity. Three different grades of postoperative fistula (grades A, B, C) are defined according to the clinical impact on the patient's hospital course.

CONTACTS AND LOCATIONS:
Overall Officials: Menghua Dai, MD, Study Director — Peking Union Medical Coll3ge hospital

IPD SHARING:
Plan to Share IPD: No